CLINICAL TRIAL: NCT04160065
Title: Phase 1 Trial of Intralesional Immunotherapy With IFx-Hu2.0 Vaccine in Patients With Advanced Non-melanoma Skin Cancers
Brief Title: Immunotherapy With IFx-Hu2.0 Vaccine for Advanced Non-melanoma Skin Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TuHURA Biosciences, Inc. (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); University of Southern California (Other); Dana-Farber Cancer Institute (Other); Huntsman Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NMSC 2019-01
Expanded Access: NCT04853602 (Available)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Merkel Cell Carcinoma; Cutaneous Squamous Cell Carcinoma; Non-Melanoma Skin Cancers
Keywords: Advanced; MCC; cSCC; pDNA; plasmid DNA; pAc/emm55; Gene Therapy; Immuno-Oncology; Therapeutic Cancer Vaccine; Immunotherapy
MeSH Terms: conditions — Carcinoma, Merkel Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IFx-Hu2.0 (plasmid DNA) 0.1 mg/lesion/time point (Experimental): Exposure Escalation:
  * The first 3 subjects enrolled will receive a fixed IFx-Hu2.0 (plasmid DNA) dose of 0.1 mg injected in up to 3 lesions at a single time point (28-day follow-up post last injection); 3/3 patients recruited.
  * The second 3 subjects enrolled will receive a fixed IFx-Hu2.0 (plasmid DNA) dose of 0.1 mg injected in up to 3 lesions at 2 time points 7 days apart (28-day follow-up post last injection); 1/3 patients recruited.
  * The third 3 subjects enrolled will receive a fixed IFx-Hu2.0 (plasmid DNA) dose of 0.1 mg injected in up to 3 lesions at 3 time points 7 days apart (28-day follow-up post last injection); recruitment pending.
  Cohort Expansion:
  * The remaining 11 subjects enrolled will receive a fixed IFx-Hu2.0 (plasmid DNA) dose of 0.1 mg injected in up to 3 lesions at 3 time points 7 days apart (28-day follow-up post last injection); recruitment pending.
  Interventions: Biological: IFx-Hu2.0

INTERVENTIONS:
Biological: IFx-Hu2.0 — The investigational drug product IFx-Hu2.0 is composed of the drug substance pAc/emm55 (pDNA) complexed with the two excipients in vivo-jetPEI® (linear polyethylenimine), a transfection reagent, and dextrose, a pDNA/polyethylenimine complex stabilizer.
  Therapeutic Classification:
  * Immunomodulatory Agent
  Route of Administration:
  * Intralesional (i.e. injection of cutaneous, subcutaneous or nodal lesions)
  Mechanism of Action:
  * Injection of IFx-Hu2.0 into the lesion facilitates the expression of the immunogenic Emm55 protein by the tumor cells.
  Physiological Effect:
  * Expression of the emm55 gene by the tumor cells triggers immune recognition of tumor-specific and -associated antigens which leads to innate and adaptive immune responses.
  Other Names: pAc/emm55

SUMMARY:
In this clinical phase I, non-randomized, open-label, uncontrolled, interventional, multi-center trial, 20 adult subjects (≥ 18 years of age) with advanced non-melanoma skin cancers will receive a fixed dose of 0.1 mg of IFx-Hu2.0 intralesionally as monotherapy in up to three lesions at up to three time points. Subjects will be observed for any acute adverse events (AEs) post injection and for any delayed AEs at Day 28, 35 and/or 42 ± 7 days, depending on the cohort (exposure escalation and expansion design).

DETAILED DESCRIPTION:
Approximately twenty adult patients (≥ 18 years of age), of any sex, ethnicity, and race with histologically confirmed advanced non-melanoma skin cancers with accessible lesions, will be eligible for study enrollment and treatment with IFx-Hu2.0 (i.e. 20 total patients across both indications). These types of advanced non-melanoma skin cancers are very rare in the pediatric population (< 18 years of age) with only scattered case reports. The potential for development of this product for pediatric subjects with non-melanoma skin cancers will be evaluated after the results of this study are available.

Patients must have at least one injectable lesion, defined as an easily palpable superficial lesion (cutaneous, subcutaneous or lymph nodal metastasis) that can be accurately localized, stabilized by palpation, and is superficial enough to enable intralesional injection.

To be eligible for this study, patients must have progressed despite standard therapy(ies), or are intolerant to or refused standard therapy(ies).

Enrollees will receive IFx-Hu2.0 as a monotherapy at up to three-time points. Depending on the number of accessible lesions, a patient could receive up to three doses across three lesions (one dose per lesion). The maximum number of lesions to be injected at any time point under this protocol is three lesions. Blood will be collected from these patients prior to treatment administration at every drug administration visit. These samples will be used to perform CBC and clinical chemistry tests. A urine sample will be obtained for urinalysis for protein and blood at the same frequency. Blood samples will also be drawn at the same intervals for immune response evaluation as well.

This is primarily a safety study that is designed to evaluate IFx-Hu2.0 monotherapy and provide foundational evidence to potentially support further studies investigating IFx-Hu2.0 + anti-PD-1 combination therapy for patients with non-melanoma skin cancers.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥ 3 months at recruitment
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at the time of study treatment initiation.
* Males or females with histologically confirmed diagnosis of advanced non-melanoma skin cancers.
* Patients must have progressed despite standard therapy(ies) or are intolerant to or refused standard therapy(ies).
* Clinically measurable disease with at least 1 injectable lesion ≥ 3 mm in longest diameter; an injectable lesion is defined as an easily palpable superficial lesion (cutaneous, subcutaneous or lymph nodal metastasis) that can be accurately localized, stabilized by palpation, and is superficial enough to enable intralesional injection.
* No known bleeding diathesis or coagulopathy that would make intratumoral injection or biopsy unsafe
* The entry laboratory criteria for subject eligibility must be less than or equal to Grade 1 adverse event levels for the parameters tested as defined by CTCAE v5.0:

  * Bone Marrow Function:

    * Hemoglobin (Hb) > LLN 10 g/dL
    * White Blood Cell Count (WBC) > LLN 3,000 cells/mcL
    * Platelet count (PLT) > LLN - 75,000 /mcL
  * Blood Coagulation Parameters

    * PT, INR < 1.5 x institutional ULN unless patient is therapeutically anticoagulated. If on anticoagulation PT/INR need to be within appropriate anticoagulation limits for the clinical indication. Patients who are receiving anticoagulants may participate in the trial if their anticoagulation can be stopped safely for several days at the time of biopsy.
  * Renal Function

    * Serum Creatinine (SCr) < 1 - 1.5 x baseline; < 1 1.5 x ULN
  * Hepatic Function:

    * Blood bilirubin < 1 - 1.5 x ULN if baseline was normal; < 1 1.5 x baseline if baseline was abnormal
    * Serum Alanine Aminotransferase (ALT) < 1 - 3 x ULN if baseline was normal; 1.5 3 x baseline if baseline was abnormal
    * Serum Aspartate Aminotransferase (AST) < 1 - 3 x ULN if baseline was normal; 1.5 3 x baseline if baseline was abnormal
    * Alkaline Phosphatase (ALP) < 1 - 2.5 x ULN if baseline was normal; 2 2.5 x baseline if baseline was abnormal
    * Gamma Glutylamyltransferase (GGT) < 1 - 2.5 x ULN, if baseline was normal; 2 2.5 x baseline if baseline was abnormal
* Males and females of reproductive potential must agree to continuously use adequate contraception prior to study entry and for up to 6 months thereafter. A female is of childbearing potential unless she has had a surgical procedure that would accomplish sterility such a bilateral tubal ligation, hysterectomy or has not had menses for the past 12 months.
* Females of childbearing potential must have a negative urine or serum pregnancy test within one week prior to start of treatment
* Patient or legal representative must understand and sign a written informed consent form.

Exclusion Criteria:

* Concurrent use of any other investigational product or participation in another trial within 28 days before start of study treatment.
* Have received oncologic therapy within 2 weeks of planned IFx-Hu2.0 injection
* Presence or history of central nervous system metastasis [treated/stable brain metastasis are allowable when patients have received prior therapy for their brain metastases and their central nervous system (CNS) disease is radiographically stable (> 4 weeks)]
* Pregnant or breastfeeding females and females desiring to become pregnant or breastfeed within the timeframe of this study
* Concurrent steroid therapy (> 10 mg of daily prednisone equivalent) or other immunosuppressive therapies such as those needed for solid organ transplants and rheumatoid arthritis. Topical or inhaled steroids are allowable.
* History of organ allograft transplantation
* History of hemolytic anemia
* History of significant tumor bleeding, or coagulation or bleeding disorders.
* Patients with autoimmune disorder, with exception of patients with vitiligo or endocrine-related autoimmune conditions receiving appropriate hormonal supplementation who are eligible; systemic use of immunosuppressant drugs such as steroids (except as hormone replacement therapy or short-course supportive medication such as chemotherapy or drug allergy, etc.), azathioprine, tacrolimus, cyclosporine, etc. within 4 weeks before recruitment. Prior autoimmune toxicity resolved to Grade 1 or less no longer requiring immunosuppressive therapy is not an exclusion under this criterion.
* Major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered major surgery) resulting from a prior surgery
* Leptomeningeal involvement regardless of treatment status
* Active, clinically serious uncontrolled medical conditions such as HIV, HBV, HCV, and EBV infection
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with protocol requirements
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Number of Grade 3-5, Treatment-Related Adverse Events per CTCAE 5.0 | 28 days from last injection

SECONDARY OUTCOMES:
Number of Enrolled Subjects who have completed the Trial without Major Protocol Deviations | 28 days from last injection
Objective Response Rate (ORR) per 2018 FDA Guidance on Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics | 28 days from last injection
Best Overall Response per RECIST v1.1 | 28 days from last injection

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Brohl, MD, Principal Investigator — Collaborator
Locations (4):
- United States (4):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No